CLINICAL TRIAL: NCT07056400
Title: Trial to Improve Fertilization Rate and Embryo Development in Intracytoplasmic Sperm Injection (ICSI) Cycles
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sci1312408001
Record Dates: First submitted 2025-06-15; First posted 2025-07-09 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-04

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- first ejaculate (Experimental): In this arm, participants will undergo ICSI using sperm collected from the first ejaculate. Semen analysis will be conducted to assess sperm quality, including motility, morphology, and concentration. This arm will serve as the baseline for comparison with the second ejaculate arm.
  Interventions: Procedure: First Ejaculate for ICSI
- Second Ejaculate (Experimental): Participants in this arm will undergo ICSI using sperm collected from the second ejaculate, which will be obtained within a short interval (1-2 hours) after the first. Semen analysis will be conducted to compare sperm quality with that of the first ejaculate, and fertilization and embryo development outcomes will be evaluated
  Interventions: Procedure: Second Ejaculate for ICSI

INTERVENTIONS:
Procedure: First Ejaculate for ICSI — Intervention 1: First Ejaculate for ICSI In this intervention, sperm collected from the first ejaculate will be used in Intracytoplasmic Sperm Injection (ICSI). The sperm will be analyzed for motility, morphology, and concentration before being used in fertilization and embryo culture. This arm will evaluate the quality of sperm obtained from the first ejaculate
  Arms: first ejaculate
Procedure: Second Ejaculate for ICSI — In this intervention, sperm collected from the second ejaculate (obtained within 1-2 hours after the first ejaculate) will be used in Intracytoplasmic Sperm Injection (ICSI). The sperm will be analyzed for motility, morphology, and concentration before being used for fertilization and embryo culture. This arm will evaluate the quality of sperm obtained from the second ejaculate and its impact on fertilization rates and embryo development
  Arms: Second Ejaculate

SUMMARY:
The Aim of the trial:

Assess if a consecutive second ejaculate contains an equal, or even higher number of motile sperm and produces high-quality sperm for intracytoplasmic sperm injection (ICSI) in male factor patients and if it will improve clinical outcomes, such as fertilization rate, embryo quality, number of blastocysts retrieved per cycle, implantation, and hopefully pregnancy rates.

DETAILED DESCRIPTION:
Background:

According to research, the length of abstinence has an impact on sperm DNA fragmentation (SDF) as well as sperm parameters. Long abstinence period increases the volume of semen and the concentration of sperm, but it will negatively impact motility, viability, and morphology.

The second ejaculation of males shows a considerable improvement in total motility and a significant decrease in (SDF) when it is collected within 1 to 3 hours of the first ejaculate.

it is essential to ensure the availability of high-quality spermatozoa with second ejaculation to enhance clinical results in ICSI cycles

ELIGIBILITY:
Inclusion Criteria:

* Male: with abnormal semen parameter according to WHO.
* Age range between 25-45 for both partners.

Exclusion Criteria:

* Female with factors that might affect Oocyte quality:

Polycystic ovary (PCO). Poor ovarian reserve. Endometriosis.

- Male partners who need testicular biopsy to retrieve sperms.

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
fertilization rate. | Periprocedural
  Fertilization will be confirmed after 16-18 hours by the observation of two distinct pronuclei (2PN) and two polar bodies. The fertilization rate will be calculated as the number of fertilized oocytes divided by total number of mature oocytes (MII) for each couple. Oocytes with 2PN will be observed

SECONDARY OUTCOMES:
Embryo development rate | periprocedural
  Oocytes with 2PN will be observed for embryonic development on day 2 and 3 until day 5 after micro-injection. The embryo development rates will be calculated as the number of embryos developed divided by the total number of mature oocytes for each couple.
semen analysis | Baseline
  Semen samples will be analyzed in both the first and second ejaculate according to the World Health Organization (WHO) 2021 guidelines. The following parameters will be assessed:
  Semen volume (mL) Sperm concentration (million/mL) Total sperm count (million) Progressive motility (%) Total motility (%) Normal morphology (%) Analysis will be performed in a certified andrology laboratory using standardized techniques.

OTHER OUTCOMES:
Clinical Pregnancy Rate | up to 6 weeks
  The clinical pregnancy rate will be assessed by detecting pregnancy via ultrasound after embryo transfer. This will help assess the long-term outcome of fertilization with sperm from the first and second ejaculates.
Sperm DNA Fragmentation index (DFI) | Baseline
  Sperm DNA fragmentation will be assessed using the HALO test (sperm chromatin dispersion assay), following the manufacturer's protocol. The DNA fragmentation index (DFI) will be calculated as the percentage of sperm cells showing fragmented DNA.

CONTACTS AND LOCATIONS:
Locations (1):
- Nour El-Hayat Fertility Center, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No